CLINICAL TRIAL: NCT01839500
Title: A Non-Interventional, Registry Study for Chinese Gastric Cancer Patients With HER2 Status: Clinical and Pathological Characteristics, Treatment Patterns and Clinical Outcomes (EVIDENCE)
Brief Title: A Non-Interventional Study of Treatment Pattern and Clinical Outcomes in Chinese Participants With Gastric Cancer
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28934
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Cohort I: HER2-Positive mGC Treated With Trastuzumab: HER2-positive metastatic gastric cancer (mGC) participants who are treated with trastuzumab will be included in this cohort. As this is an observational study, treatment schedule will be at the clinician's discretion in accordance with routine care practice and not dictated by the protocol.
  Interventions: Drug: Trastuzumab
- Cohort II: HER2-Positive mGC not Treated With Trastuzumab: HER2-positive mGC participants who are not treated with trastuzumab will be included in this cohort.
- Cohort III: HER2-Positive non-mGC: HER2-positive non-mGC participants will be included in this cohort.
- Cohort IV: HER2-Negative mGC: HER2-negative mGC participants will be included in this cohort.
- Cohort V: HER2-Negative non-mGC: HER2-negative non-mGC participants will be included in this cohort.

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab administered in accordance with routine care practice.
  Other Names: Herceptin
  Groups: Cohort I: HER2-Positive mGC Treated With Trastuzumab

SUMMARY:
This prospective, multi-center, non-interventional study will evaluate the efficacy and safety of trastuzumab in routine clinical practice in Chinese participants with gastric or gastro-oesophageal cancer. The study will be conducted in 5 cohorts and eligible participants will be enrolled and assigned to the various cohorts according to human epidermal growth factor receptor 2 (HER2) status, disease stage and treatment with trastuzumab according to physician's decision. Treatment patterns and clinical outcomes in participants with gastric cancer in China will be evaluated. The total study duration is 60 months.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Histologically confirmed cancer of the stomach or gastro-oesophageal junction or recurrent disease within 6 months before the date of recruitment
* Documented participant with trackable medical records
* HER2 status by immunohistochemistry (IHC) is known

Specific Inclusion Criteria:

* Cohort I/II/IV: Participants with mGC: with recurrent or metastatic disease or with inoperable locally advanced disease
* Cohort III/V: Participants with operable non-mGC: TxNxM0 (according to American Joint Committee on Cancer [AJCC] edition 7th)

Exclusion Criteria:

* Participants receiving regimen in a blinded trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with gastric or gastro-oesophageal junction cancers in China
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2013-04-25 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Baseline up to death (up to approximately 5 years)
Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR), as Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1) Criteria | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
Cohort I, II, IV: Time to Treatment Failure (TTF), as Assessed by the Investigator Using RECIST V1.1 Criteria | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
Cohort I, II, IV: Progression-Free Survival (PFS), as Assessed by the Investigator Using RECIST V1.1 Criteria | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)
Cohort III, V: Event-Free Survival (EFS), as Assessed by the Investigator Using RECIST V1.1 Criteria | Baseline up to disease recurrence or progression or death, whichever occurs first (up to approximately 5 years)
Cohort III, V: Disease-Free Survival (DFS), as Assessed by the Investigator Using RECIST V1.1 Criteria | Baseline up to disease progression or death, whichever occurs first (up to approximately 5 years)

SECONDARY OUTCOMES:
Cohort I: Percentage of Participants With Non-Serious Adverse Events and Serious Adverse Events | Baseline up to approximately 5 years
Percentage of Participants Treated with Various Initial and Subsequent Therapies (Chemotherapy, Targeted, or Investigational Treatments) | Baseline up to approximately 5 years
Cohort II: Percentage of Healthcare Professionals (HCPs) Who Recommend Treatment According to Guideline | Baseline up to first follow-up (up to approximately 5 years)
Cohort II: Percentage of Participants Who Decline to the Recommendation Categorized by Reasons | Baseline up to first follow-up (up to approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (81):
- China (81):
  - Anyang Tumor Hosptial, Anyang
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Peking University First Hospital, Beijing
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - the First Hospital of Jilin University, Changchun
  - Hu Nan Provincial Cancer Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Changzhou First People's Hospital, Changzhou
  - Sichuan Provincial Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - Fujian Medical University Union Hospital, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Fujian Provincial Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - Guizhou Cancer Hospital, Guiyang
  - Hainan provincial people's hospital, Haikou
  - Cancer Hospital of Hangzhou (Wushan District), Hangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Inner Mongolia People's Hospital, Hohhot
  - Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - The First Affilliated Hospital of Kunming Medical College, Kunming
  - The First People's Hospital of Yunnan Province, Kunming
  - Yunnan Cancer Hospital, Kunming
  - The First Affiliated Hospital of Lanzhou University, Lanzhou
  - Gansu Cancer Hospital, Lanzhou
  - Taizhou Hospital of Zhejiang Province, Linhai
  - The First Affiliated Hospital of Henan UN of Science and Technology, Luoyang
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Jiangxi Cancer Hospital; First department of abdominal surgery, Nanchang
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Nanjing 1st Hospital; Endocrinology Dept., Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The 81st Hospital of P.L.A., Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Nan Tong Tumor Hospital, Nantong
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Changhai Hospital of Shanghai, Shanghai
  - Changhai Hospital; Oncology, Shanghai
  - Shaoxing People's Hospital, Shaoxing
  - Liaoning cancer Hospital & Institute, Shenyang
  - Hebei Medical University Fourth Hospital;(Tumor Hospital of Hebei Province), Shijiazhuang
  - First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Province Cancer Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin (天津)
  - The Tumor Hospital of Xinjiang Medical University, Ürümqi
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi
  - The Second Affiliated Hospital & Yuying Children's Hospital of Wenzhou Medical College, Wenzhou
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Wuxi No.4 People's Hospital, Wuxi
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - Shanxi Provincial People's Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Xiamen University, Xiamen
  - Xinxiang Central Hospital, Xinxiang
  - Northern Jangsu People's Hospital, Yangzhou
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang